CLINICAL TRIAL: NCT04209725
Title: A Phase II Study Assessing CPX-351 (Vyxeos™) With Quizartinib for the Treatment of Relapsed or Refractory FLT3-ITD Mutation-Positive AML
Brief Title: A Study of CPX-351 (Vyxeos™) With Quizartinib for the Treatment of FLT3-ITD Mutation-Positive Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed due to slow enrollment
Sponsor: SCRI Development Innovations, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI AML 48
Record Dates: First submitted 2019-12-20; First posted 2019-12-24 (Actual); Results first posted 2022-06-03 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2022-05

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: FLT3
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — CPX-351; quizartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CPX-351 and Quizartinib treatment (Experimental): Participants with FLT3 mutation positive AML will be given CPX-351 followed by quizartinib in three phases: induction, consolidation, and maintenance.
  Interventions: Drug: CPX-351; Drug: Quizartinib

INTERVENTIONS:
Drug: CPX-351 — Given during the induction and consildation phase and will consist of 44 mg/m^2 daunorubicin with 100 mg/m^2 cytarabine administered intravenously on Days 1, 3, and 5 during induction phase and Days 1 and 3 of consolidation phase.
  Other Names: Vyxeos
Drug: Quizartinib — Given during induction, consolidation, and maintenance phases and will be taken orally at a dose of 30mg on Days 8-21 of induction phase, Days 6-21 of consolidation phase, and daily in maintenance phase.

SUMMARY:
This is a research study to be done at multiple sites in participants with advanced acute myeloid leukemia (AML) that have a mutation in Fms-like tyrosine kinase-3 internal tandem duplications (FLT3-ITD). This study is to learn more about an investigational drug, quizartinib, being tested with the anti-cancer medicine CPX-351 (also called Vyxeos™), which is approved and widely used to treat AML.

The purpose of this study is to assess the safety, tolerability and survival of patients receiving the combination of CPX-351 and quizartinib.

DETAILED DESCRIPTION:
This is an open-label, two-part Phase II clinical trial in patients with relapsed or refractory FLT3-ITD mutation-positive acute myeloid leukemia (AML). The study is designed to assess the safety and tolerability as well as the efficacy of administering CPX-351 (cytarabine:daunorubicin liposome complex) with quizartinib. CPX-351 is a formulation of two drugs, cytarabine and daunorubicin, that is administered as the first part of treatment to get rid of as many leukemia cells in your bone marrow as possible. Quizartinib is an investigational drug made of a protein that inhibits FLT3 and will be given after CPX-351 has been given. The plan for administration is divided into three phases: induction, consolidation, and maintenance.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent form (ICF), according to local guidelines, signed by the patient or by a legal guardian prior to the performance of any study-related screening procedures.
2. Patients with the following types of AML with >5% blasts:

   * Relapsed FLT3-ITD mutation-positive AML, diagnosed by bone marrow (BM) biopsy with FLT3 mutation by polymerase chain reaction (PCR)
   * Refractory FLT3-ITD mutation-positive AML, diagnosed by BM biopsy with FLT3 mutation by PCR
   * Relapsed or refractory FLT3-ITD mutation-positive AML after HCT, diagnosed by BM biopsy with FLT3 mutation by PCR
   * Relapsed or refractory AML with de novo FLT3-ITD mutation, diagnosed by BM biopsy with FLT3 mutation by PCR
   * Relapsed or refractory AML after HCT with de novo FLT3-ITD mutation, diagnosed by BM biopsy with FLT3 mutation by PCR
3. First-line therapy must have contained a standard induction chemotherapy (e.g. 7+3, FLAG-IDA, FLAG, CLAG, MEC, hypomethylating agent with venetoclax) with or without receiving a prior FLT3 inhibitor (e.g. midostaurin) or multi-tyrosine kinase inhibitor (e.g. sorafenib). All patients who relapsed after an alloHCT are included, except patients with active graft-versus-host disease (GVHD) requiring >10 mg prednisone.
4. Patients must be able to swallow and retain oral medication.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0, 1, or 2 (Appendix A).
6. Adequate renal and hepatic parameters (aspartate aminotransferase [AST], alanine aminotransferase [ALT] ≤2.5 institutional upper limit of normal [ULN]; total bilirubin ≤2.0 institutional ULN; serum creatinine [Cr] ≤2.0). In patients with suspected liver infiltration, ALT can be ≤5 institutional ULN.

Exclusion Criteria:

1. Acute promyelocytic leukemia (t[15;17])
2. Female patients who are lactating or have a positive serum pregnancy test during the screening period. Female patients of childbearing potential who are not willing to employ highly effective birth control (as defined in Appendix C of protocol) from screening to 6 months following the last dose of CPX-351 and/or quizartinib.
3. Evidence of active and uncontrolled bacterial, fungal, parasitic, or viral infection. Infections are considered controlled if appropriate therapy has been instituted and, at the time of screening, no signs of active infection progression are present. This is assessed by the site clinicians, including an infectious disease consulting physician, if requested by the Principal Investigator (PI), regarding adequacy of therapy. These infections include, but are not limited to:

   * Known human immunodeficiency virus (HIV) infection
   * Active hepatitis B or C infection with rising transaminase values
   * Active tuberculosis infection
4. History of hypersensitivity to cytarabine, daunorubicin, or an FLT3 inhibitor
5. Any patients with known significant impairment in gastrointestinal (GI) function or GI disease that my significantly alter the absorption of quizartinib.
6. Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
7. Uncontrolled or significant cardiovascular disease, including any of the following:

   * Bradycardia of less than 50 beats per minute, unless the patient has a pacemaker
   * QTcF interval using Fridericia's correction factor (QTcF) interval prolongation, defined as >450msec at screening and prior to first administration of quizartinib
   * Diagnosis of or suspicion of long QT syndrome (including family history of long QT syndrome)
   * Systolic blood pressure ≥180 mmHg or diastolic blood pressure ≥110 mmHg
   * History of clinically relevant ventricular arrhythmias (i.e., ventricular tachycardia, ventricular fibrillation or Torsades de pointes)
   * History of second or third degree heart block without a pacemaker
   * Right bundle branch and left anterior hemiblock (bifascicular block), complete left bundle branch block
   * Ejection fraction <50% by transthoracic echocardiogram (TTE) or multigated acquisition (MUGA) scan
   * History of uncontrolled angina pectoris or myocardial infarction within 6 months prior to Screening
8. History of New York Heart Association Class 3 or 4 heart failure
9. Prior anthracycline (or equivalent) cumulative exposure ≥368 mg/m2 daunorubicin (or equivalent)
10. Any serious underlying medical condition that, in the opinion of the Investigator or Medical Monitor, would impair the ability to receive or tolerate the planned treatment.
11. Patients with inadequate adequate pulmonary function will be excluded. Inadequate pulmonary function is defined as requiring supplemental O2, or diffusing capacity of the lungs for carbon monoxide [DLCO] <40%.
12. Active acute or chronic GVHD requiring prednisone >10 mg or equivalent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Tees, MD, MPH, Study Chair — Colorado Blood Cancer Institute
Locations (5):
- United States (5):
  - Colorado Blood Cancer Institute, Denver, Colorado
  - HCA Midwest, Kansas City, Missouri
  - Tennessee Oncology, Nashville, Tennessee
  - St. David's South Austin Medical Center, Austin, Texas
  - Texas Transplant Institute, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- CPX-351 and Quizartinib Treatment: Participants with FLT3 mutation positive AML will be given CPX-351 followed by quizartinib in three phases: induction, consolidation, and maintenance. CPX-351: To be given during the induction and consolidation phase and will consist of 44 mg/m^2 daunorubicin with 100 mg/m^2 cytarabine administered intravenously on Days 1, 3, and 5 during induction phase and Days 1 and 3 of consolidation phase. Quizartinib: To be given during induction, consolidation, and maintenance phases and will be taken orally at a dose of 30mg on Days 8-21 of induction phase, Days 6-21 of consolidation phase, and daily in maintenance phase.
Period: Overall Study
Arm/Group | CPX-351 and Quizartinib Treatment
Started | 1
Completed | 0
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Only 1 patient was enrolled and treated before study was terminated due to slow accrual
Arm/Group | CPX-351 and Quizartinib Treatment
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Treatment Related Adverse Events After Taking CPX-351 and Quizartinib
Description: Counting the number of patients with treatment related adverse events as a measure of safety and tolerability.
Time Frame: Collected during treatment and for 30 days after last dose, approximately 35 total days for the 1 patient treated.
Population: 1 patient was treated on study and did have treatment-related adverse events
Measure: Count of Participants; unit: Participants
Arm/Group | CPX-351 and Quizartinib Treatment
Number analyzed (Participants) | 1
Participants | 1

2. Primary Outcome: Number of Patients With an Overall Response Taking CPX-351 and Quizartinib
Description: Overall response is defined by the International Working Group response criteria (Cheson et al 2003) as having a complete remission (CR) - a complete morphologic response with complete blood count recovery absolute neutrophil count ≥1000/μL and platelet count ≥100,000/μL) or a complete morphologic response with an incomplete blood count recovery (CRi) - absolute neutrophil count <1000/μL and/or platelet count <100,000/μL)
Time Frame: from cycle 1 day 1 (each cycle is 28 days) until disease progression for up to 2 years post treatment
Population: Patients must have received at least one dose of CPX-351 or quizartinib, who have an adequate baseline disease assessment, and an adequate post-baseline assessment and who discontinue due to death or PD prior to their first assessment. The 1 patient that was enrolled discontinued study treatment in Cycle 1 prior to receiving Quizartinib, no post-baseline assessment was done. Therefore, no patients were analyzed.
Arm/Group | CPX-351 and Quizartinib Treatment
Number analyzed (Participants) | 0

3. Secondary Outcome: Median Time to Platelet Count Recovery
Description: Time to platelet recovery is defined as the time to when the peripheral blood platelet count is >50, 000/ μL
Time Frame: from cycle 1 Day 1 (each cycle is 28 days) for up to 24 months
Population: The 1 patient that was enrolled discontinued study treatment in Cycle 1 prior to receiving Quizartinib, no post-baseline assessment was done. Therefore, no patients were analyzed.
Arm/Group | CPX-351 and Quizartinib Treatment
Number analyzed (Participants) | 0

4. Secondary Outcome: Median Time to Absolute Neutrophil Count (ANC) Recovery
Description: Time to neutrophil recovery is defined as the time to when the peripheral blood ANC is ≥500/μL
Time Frame: from Cycle 1 Day 1 (each cycle is 28 days) for up to 24 months
Population: as for outcome 3
Arm/Group | CPX-351 and Quizartinib Treatment
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Patients Proceeding to an Allogeneic Hematopoietic Cell Transplantation (alloHCT)
Description: Patients receiving allogeneic hematopoietic cell transplantation (alloHCT) following treatment in induction and consolidation therapies.
Time Frame: up to 60 days after consolidation therapy
Population: The patient discontinued treatment early and didn't follow induction and consolidation therapies to reach the alloHCT. Therefore no patients were analyzed.
Arm/Group | CPX-351 and Quizartinib Treatment
Number analyzed (Participants) | 0

6. Secondary Outcome: Median Time to Disease Progression
Description: Time to disease progression, confirmed by bone marrow biopsy.
Time Frame: from diagnosis of relapse or refractory AML until disease progression for up to 2 years post treatment
Population: The 1 patient that was enrolled discontinued study treatment in Cycle 1 prior to receiving Quizartinib, no post-baseline evaluation was done. Therefore, no patients were analyzed.
Arm/Group | CPX-351 and Quizartinib Treatment
Number analyzed (Participants) | 0

7. Secondary Outcome: Event-free Survival Time
Description: Defined as the number of days until evidence of PD by bone marrow biopsy/aspirate, or death, regardless of cause. Patients who are alive without a disease response assessment of relapsed disease will be censored at the last adequate disease assessment date. Patients without a disease response assessment will be censored at the first date of treatment.
Time Frame: from day 1 for up to 4 years
Population: The 1 patient that was enrolled discontinued study treatment in Cycle 1 prior to receiving Quizartinib. No post-baseline assessment was performed and was therefore censored at Date of First Treatment. Therefore, no patients were analyzed.
Arm/Group | CPX-351 and Quizartinib Treatment
Number analyzed (Participants) | 0

8. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from the first date of treatment until death as a result of any cause. For OS time, patients that have not died or are lost to follow-up will be censored at the date the patient was last known to be alive or the date of last contact.
Time Frame: Up to 8 months
Population: Only 1 patient was treated.
Measure: Number; unit: months
Arm/Group | CPX-351 and Quizartinib Treatment
Number analyzed (Participants) | 1
months | 7.7

9. Secondary Outcome: Number of Patients Who Develop Late Responses
Description: Late responses as defined by the International Working Group response criteria (Cheson et al 2003) as having a complete remission (CR) - a complete morphologic response with complete blood count recovery absolute neutrophil count ≥1000/μL and platelet count ≥100,000/μL) or a complete morphologic response with an incomplete blood count recovery (CRi) - absolute neutrophil count <1000/μL and/or platelet count <100,000/μL
Time Frame: up to 4 years
Population: as for outcome 3
Arm/Group | CPX-351 and Quizartinib Treatment
Number analyzed (Participants) | 0

10. Secondary Outcome: Number of Patients Who Can Receive Consolidation and Maintenance Therapy
Description: Patients who proceed through induction to next stages of consolidation and maintenance
Time Frame: approximately 3 months
Population: The patient discontinued treatment early and didn't follow induction and consolidation therapies to reach the alloHCT or maintenance therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | CPX-351 and Quizartinib Treatment
Number analyzed (Participants) | 1
Participants | 0

11. Secondary Outcome: Treatment-related Mortality Rate
Description: As determined by the number of treatment related deaths during study treatment
Time Frame: Observed during treatment and for 30 days after last dose, so approximately 35 days for the 1 patient treated.
Population: The 1 enrolled patient did not have a treatment-related death.
Measure: Count of Participants; unit: Participants
Arm/Group | CPX-351 and Quizartinib Treatment
Number analyzed (Participants) | 1
Participants | 0

12. Secondary Outcome: Percentage of Patients Who Achieve a PR or Molecular Complete Remission
Description: A PR is defined as persistent disease by morphology but with a >50% reduction in the blast count/cellularity ratio compared to the most recent BM biopsy prior to treatment. A molecular complete remission is defined as no evidence of disease by bone marrow biopsy/aspirate by morphology, immunohistochemistry, or flow cytometry, and FLT3 mutation by MRD analysis.
Time Frame: from cycle 1 day 1 (each cycle is 28 days) until disease progression for up to 2 years post treatment
Population: as for outcome 3
Arm/Group | CPX-351 and Quizartinib Treatment
Number analyzed (Participants) | 0

13. Secondary Outcome: Mean Elapsed Time for Patients to Achieve Molecular CR
Description: The mean time to achievement of a complete morphologic CR with persistent disease detected by flow or molecular minimal residual disease (MRD) analysis.
Time Frame: From Date of First Treatment to up to 2 years
Population: The 1 patient enrolled discontinued in Cycle 1. No post-baseline assessment therefore no patients analyzed
Arm/Group | CPX-351 and Quizartinib Treatment
Number analyzed (Participants) | 0

14. Secondary Outcome: Quizartinib Tolerability After Allogeneic Hematopoietic Cell Transplantation (alloHCT) or Donor Lymphocyte Infusion (DLI)
Description: Defined as the number of patients who received quizartinib and proceeded to alloHCT or DLI as part of this study and had treatment-related adverse events
Time Frame: From Date of First Treatment, up to 2 years
Population: The 1 patient enrolled discontinued the study prior to receiving their first dose of quizartinib. Therefore no patients analyzed.
Arm/Group | CPX-351 and Quizartinib Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Collected for 30 days after last dose, so approximately 35 days for the 1 patient treated.
Description: All patients who received at least one dose of protocol treatment were followed for safety. Adverse events and serious adverse events were collected from day of first dose to 30 days after last protocol treatment and graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Arm/Group | CPX-351 and Quizartinib Treatment
All-Cause Mortality (participants affected / at risk) | 1/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CPX-351 and Quizartinib Treatment (N=1)
Anaemia (Blood and lymphatic system disorders) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-10): https://cdn.clinicaltrials.gov/large-docs/25/NCT04209725/Prot_SAP_000.pdf